CLINICAL TRIAL: NCT01938222
Title: A Prospective, Controlled Monocentric Study Evaluating the 6:1 Suture Technique Using Suture Material Monomax® for Abdominal Wall Closure After Primary Abdominal Incision
Brief Title: Short Stitch Monomax®
Acronym: Short-Stitch
Status: Completed | Type: Observational
Sponsor: Diakonie-Klinikum Schwäbisch Hall gGmbH (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-I-H-1203
Record Dates: First submitted 2013-08-26; First posted 2013-09-10 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Dehiscence of Laparotomy Wound; Surgical Wound Infection
Keywords: abdominal wall closure; short stitch technique
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Short Stitch: Short stitch suture technique (6:1) for abdominal all closure stitch interval < 0,5 cm and lateral 0,5-0,8 cm
  Interventions: Procedure: Short Stitch

INTERVENTIONS:
Procedure: Short Stitch — MonoMax® suture material USP (United States Pharmacopeia) 2/0, 150 cm, HR (half-round) 26 mm needle, will be applied in the short stitch technique (6:1) for abdominal wall closure.
  Other Names: MonoMax®

SUMMARY:
A number of studies identifies abdominal hernia as the most frequent postoperative complication following laparotomy with percentages of 9-20% - depending on duration of follow-up. It is based on a multifactorial basis, including factors concerning individual, patient-specific factors, factors related to the operational technique as well as particular surgical factors. Wound complications have been reported by 7-12%, burst abdomen rate (dehiscence) < 5 days being 2-4%, wound infection rate (+/- wound dehiscence) ≥ 5 days being 6-10%. In emergency procedures (e.g. ileus, perforation of hollow organ) a wound complication rate of up to 50 % has to be expected. According to new, first findings from recent studies the rates of wound healing complication and burst abdomen can be reduced significantly. Depending on the study, to almost 50%. The principle is based on the reduction of the stitch length and type of the inserted suture. The stitches are closer and with less distance to the edge of fascia. Due to the much thinner suture it still comes here to a quantitative reduction of the inserted suture. The data collected using the MonoMax® suture in the short stitch technique will be compared to the results of the ISSAAC trial, in which the MonoMax® suture was used in the long stitch suture technique. The generated data are thus subject of retrospective comparison with a historical control group (ISSAAC study).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Primary elective and primary emergency laparotomy
* Written informed consent

Exclusion Criteria:

- Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Wound-infection rate until day of discharge according to CDC (Centre of Disease Control) Classification | until discharge (ca. 10 days after operation)

SECONDARY OUTCOMES:
Reoperation rate due to burst abdomen until discharge | until discharge (ca. 10 days after operation)
Wound healing complications until discharge | until discharge (ca. 10 days after operation)
Length of postoperative hospital stay | until discharge (ca. 10 days after operation)
Use of the suture material (tissue drag, elasticity, knot security, knot pull tensile strength, knot run-down) | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Markus Golling, Prof., Principal Investigator — Diakonie-Klinikum Schwäbisch Hall gGmbH
Locations (1):
- Diakonie Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall, Germany

REFERENCES:
- [Background] Golling M, Breul V, Zielska Z et al. 6:1 Suture or Wound length ratio with the short stitch technique - a reality check on practicability and short term outcome. Sur Res J. 2022;2(2).
- [Result] Golling M, Breul V, Zielska Z, Baumann P. The 6:1 short stitch SL-WL-ratio: short term closure results of transverse and midline incisions in elective and emergency operations. Hernia. 2024 Apr;28(2):447-456. doi: 10.1007/s10029-023-02927-4. Epub 2024 Jan 29. PMID 38285168